CLINICAL TRIAL: NCT00988039
Title: A Randomised Controlled Trial to Evaluate Options for Second-line Therapy in Patients Failing a First-line 2NRTI + NNRTI Regimen in Africa
Brief Title: Europe-Africa Research Network for Evaluation of Second-line Therapy
Acronym: EARNEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Justine Boles (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor-Investigator, Justine Boles, Professor Nicholas Paton, Medical Research Council
Organization: Medical Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U.1228.03.004.00021.01; IP_2007_33011_003; ISRCTN37737787
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Human Immunodeficiency Virus; HIV
Keywords: Human Immunodeficiency virus; second line therapy; raltegravir; aluvia; monotherapy; integrase inhibitor; protease inhibitor; Randomized Controlled Trial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — lopinavir-ritonavir drug combination; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- bPI + 2NRTIs (Active Comparator)
  Interventions: Drug: Aluvia + 2NRTIs
- bPI + raltegravir (Experimental)
  Interventions: Drug: Aluvia + raltegravir
- bPI monotherapy (Experimental)
  Interventions: Drug: Aluvia monotherapy

INTERVENTIONS:
Drug: Aluvia + 2NRTIs — Aluvia (lopinavir/ritonavir 400mg/100mg), twice daily
  The choice of NRTIs will be at the discretion of the managing clinician and based on the local standard of care and drug availability, taking into account patient's previous drug exposure and side effects on first-line therapy.
  Arms: bPI + 2NRTIs
Drug: Aluvia + raltegravir — Aluvia (lopinavir/ritonavir 400mg/100mg) twice daily
  raltegravir (400mg) twice daily
  Arms: bPI + raltegravir
Drug: Aluvia monotherapy — Aluvia (lopinavir/ritonavir 400mg/100mg) twice daily
  raltegravir (400mg) twice daily for the first 12 weeks only
  Arms: bPI monotherapy

SUMMARY:
The trial aim is to ascertain what, if anything, needs to be combined with a boosted protease inhibitor (bPI) backbone in second-line therapy in order to maximize the chance of a good clinical outcome following WHO-defined failure on a first-line nucleoside reverse transcriptase inhibitor (NRTI) and NNRTI-containing regimen with probable extensive NRTI and NNRTI resistance mutations.

DETAILED DESCRIPTION:
The standard of care for second-line HIV therapy in patients who have failed a first-line NNRTI-based regimen is to combine a boosted protease inhibitor (bPI) with two (new) NRTIs. However, patients failing first-line therapy in roll-out programmes often have extensive NRTI resistance mutations that may compromise the efficacy of the NRTI drugs used in second-line therapy and it is likely that the virological potency of the second-line regimen is mostly due to the bPI. It is possible that the contribution of the NRTI drugs to efficacy may be outweighed by additional toxicity and cost. It is also possible that replacing the NRTI drugs with a new class of drug (integrase inhibitors) will improve outcome from second-line therapy, although if the boosted protease inhibitor alone is providing close to optimal response, incremental gains from adding a new class may be small.

The principal aims are to determine whether, in patients failing a first-line NRTI and NNRTI-containing regimen:

* The use of bPI plus raltegravir (an integrase inhibitor) is superior to standard of care (bPI plus 2 new NRTIs) in achieving good HIV disease control at 96 weeks after randomisation
* The use of bPI monotherapy, preceded by a 12-week induction period in combination with raltegravir, is non-inferior to standard of care in achieving good HIV disease control at 96 weeks after randomisation

ELIGIBILITY:
Inclusion Criteria:

* Previously documented HIV infection on at least one standard antibody-based test
* Age 12 years and above
* Taking 2NRTI + NNRTI-based regimen continuously for at least 12 months
* Naive to protease inhibitor therapy
* Good adherence to ART in the 12 weeks prior to screening defined as missing medication on no more than 3 days in the prior month
* Clinically stable and receiving treatment for any known opportunistic infections
* HIV treatment failure defined by one or more of clinical, immunological or virological criteria defined in the protocol, including VL and CD4 at screening visit
* Willing and able to give informed consent
* Able to attend for regular study follow up visits

Exclusion Criteria:

* Any major clinical contra-indications to the use of bPI, the NRTIs that are available to be selected for a second-line regimen or raltegravir
* Known Hepatitis B carrier (Hepatitis B surface antigen positive if tested)
* Requires concomitant medication with known major interactions with study drugs for which drug substitutions or dose alterations are not available or acceptable
* Women who are currently pregnant or breastfeeding
* Current participation in another clinical trial involving a treatment intervention (may be permitted in some circumstances, but must be discussed with MRC CTU)
* Life expectancy of less than one month in the opinion of the treating physician

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1277 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Good HIV disease control defined as a composite endpoint consisting of all of: - No new WHO stage 4 events - CD4 count >250 cells/mm3 - viral load <10,000 copies/ml or >10,000 copies/ml with no PI resistance mutations | week 96

SECONDARY OUTCOMES:
Good HIV disease control | week 144
Proportion with CD4 cell count >250 cells/mm3 | week 96 and week 144
Proportion with new or recurrent WHO stage 4 event | week 96 and week 144
Proportion of patients with plasma viral load <50 copies | week 48, week 96 and week 144
Adverse events | During trial
Quality of life change from randomisation | During trial
Neurocognitive function change from randomisation | during trial
Healthcare costs | During trial
Proportion with serious non-AIDS events | Week 96 and week 144

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, MD FRCP, Study Director — MRC CTU
Locations (14):
- AMPATH Centre at Moi Teaching Referral Hospital, Eldoret, Kenya
- Malawi (2):
  - University of Malawi, Blantyre
  - Mzuzu Central Hospital, Mzuzu
- Uganda (9):
  - Joint Clinical Research Centre, Fort Portal
  - JCRC, Gulu
  - JCRC, Kabale
  - JCRC, Kakira
  - Infectious Diseases Institute, Kampala
  - Joint Clinical Research Centre, Kampala
  - San Raphael of St Francis Hospital Nsambya, Kampala
  - Joint Clinical Research Centre, Mbale
  - Joint Clinical Research Centre, Mbarara
- University Teaching Hospital, Lusaka, Zambia
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

REFERENCES:
- [Derived] Shi Y, Thompson J, Walker AS, Paton NI, Cheung YB; EARNEST Trial Team. Mapping the medical outcomes study HIV health survey (MOS-HIV) to the EuroQoL 5 Dimension (EQ-5D-3 L) utility index. Health Qual Life Outcomes. 2019 May 10;17(1):83. doi: 10.1186/s12955-019-1135-8. PMID 31077251
- [Derived] Thompson JA, Kityo C, Dunn D, Hoppe A, Ndashimye E, Hakim J, Kambugu A, van Oosterhout JJ, Arribas J, Mugyenyi P, Walker AS, Paton NI; Europe-Africa Research Network for Evaluation of Second-line Therapy (EARNEST) Trial Team. Evolution of Protease Inhibitor Resistance in Human Immunodeficiency Virus Type 1 Infected Patients Failing Protease Inhibitor Monotherapy as Second-line Therapy in Low-income Countries: An Observational Analysis Within the EARNEST Randomized Trial. Clin Infect Dis. 2019 Mar 19;68(7):1184-1192. doi: 10.1093/cid/ciy589. PMID 30060027
- [Derived] Paton NI, Kityo C, Thompson J, Nankya I, Bagenda L, Hoppe A, Hakim J, Kambugu A, van Oosterhout JJ, Kiconco M, Bertagnolio S, Easterbrook PJ, Mugyenyi P, Walker AS; Europe Africa Research Network for Evaluation of Second-line Therapy (EARNEST) Trial Team. Nucleoside reverse-transcriptase inhibitor cross-resistance and outcomes from second-line antiretroviral therapy in the public health approach: an observational analysis within the randomised, open-label, EARNEST trial. Lancet HIV. 2017 Aug;4(8):e341-e348. doi: 10.1016/S2352-3018(17)30065-6. Epub 2017 May 8. PMID 28495562
- [Derived] Paton NI, Kityo C, Hoppe A, Reid A, Kambugu A, Lugemwa A, van Oosterhout JJ, Kiconco M, Siika A, Mwebaze R, Abwola M, Abongomera G, Mweemba A, Alima H, Atwongyeire D, Nyirenda R, Boles J, Thompson J, Tumukunde D, Chidziva E, Mambule I, Arribas JR, Easterbrook PJ, Hakim J, Walker AS, Mugyenyi P; EARNEST Trial Team. Assessment of second-line antiretroviral regimens for HIV therapy in Africa. N Engl J Med. 2014 Jul 17;371(3):234-47. doi: 10.1056/NEJMoa1311274. PMID 25014688
- See also: EARNEST trial website — http://earnest.cineca.org/